CLINICAL TRIAL: NCT06339606
Title: Repository for Biospecimens From Pregnant Patients
Brief Title: Pregnancy Repository
Acronym: PR
Status: Not yet recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 4316
Record Dates: First submitted 2024-03-15; First posted 2024-04-01 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy Related; Fetal Growth Retardation; Placental Insufficiency; Preeclampsia; Cervix; Pregnancy
MeSH Terms: conditions — Fetal Growth Retardation; Placental Insufficiency; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples With DNA — Blood samples (up to 20 mL) will be collected serially during pregnancy. Cervical swabs will be collected serially during the first 30 weeks of pregnancy.
  Tissue specimens from the placenta (1-5 g) will be collected after delivery. Umbilical cord blood (10 mL) will be collected after delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Abnormal Placentation: Women with a singleton or multiple pregnancy that are known or suspected of having abnormal placentation
  Interventions: Other: Biospecimen collection
- Control: Women with a singleton or multiple pregnancy with a low-risk pregnancy.
  Interventions: Other: Biospecimen collection

INTERVENTIONS:
Other: Biospecimen collection — Biospecimens, including maternal blood and cervical mucus will be collected serially during pregnancy. After delivery tissue samples from the placenta and umbilical cord blood will be collected.
  Other Names: Registry/data collection from subject's medical records

SUMMARY:
An essential part of clinical research is the availability and accessibility of human biospecimens for the identification of biomarkers, new treatments and measurement of response to therapy. Proteins, RNA and DNA can be extracted and studied as well. This is a critical first step in performing many fundamental molecular biology experiments. A variety of biospecimens are utilized for research including but not limited to normal and malignant tissues, blood, and other body fluids.

In order to obtain high-quality biospecimens, they must be acquired serially, stored according to current standards, and matched with clinical information for maximum value. As such, the investigators would like to create a repository of biospecimens collected from pregnant patients who are seen at Mount Sinai Hospital and other research hospitals in Toronto. Mount Sinai provides personnel and infrastructure to serve the largest (7500 births/year) and highest complex Maternity program in Ontario. Of the 7500 patients a year, at least 2500 are considered high risk pregnancies, where there's a possibility of preeclampsia, placenta accreta and a host of other complications. For this study, biological specimens - blood, cervical and placental samples - will be collected from these high-risk groups in order to better understand the causes of the underlying conditions.

DETAILED DESCRIPTION:
The study will be non-interventional and designed for prospective sample collection and concurrent analysis.

Primary Objective #1: The primary objective is to provide a mechanism for system-wide patient engagement for banking and sourcing high-quality biologic specimens including tissues and bodily fluids. The study will be initiated at 3 sites - Sunnybrook Health Sciences Centre, North York General Hospital and Mt.Sinai Hospital - in the hopes of creating a translational research environment where patient data and biospecimens can inform future clinical practice.

The aim is to do this by:

1. Establishing a comprehensive, secure and de-identified registry/database that includes current and future cases at high risk for abnormal placentation and healthy controls for comparison with patient consent.
2. Comparing cases of suspected abnormal placentation with a control group of women with no evidence of abnormal placentation.

Primary Objective #2: Feasibility study that aims to provide preliminary insights into the biological markers and processes associated with abnormal placentation. By comparing a larger control group to those experiencing abnormal placentation, the investigators seek to understand potential biomarker differences. This phase is explorative in nature and is designed to determine the viability of our research approach and generate preliminary data.

Secondary Objective: The secondary objective is to facilitate research studies with utilization of these biologic specimens, including full-scale trials, should our initial findings warrant them.

The blood samples will be useful in identifying the molecular biomarkers that are indicative of disease, while the placental and cervical samples are important to better understand the underlying physiology of perinatal disease. The aim is therefore to establish both a clinical database and a blood/tissue bio-bank. By more comprehensively understanding the pathophysiology of invasive placentation, the goal is to develop high specificity testing modalities, perhaps through novel maternal serum biomarkers, to aid in diagnosis, management and improved outcomes for both mothers and their babies.

Patients will be consented during their visit to the hospital, and blood/cervical samples will be collected serially at each visit. Patient data will be collected from the Electronic Medical Record systems and paper charts, and this will be entered into REDCap. The biological samples will be sent to Sunnybrook Research Institute for storage.

Both blood and tissue specimens will be collected during regular patient visits. Biospecimens will be labeled with an anonymous study identifier that will be linked to corresponding clinical data and specimen annotation. Specimens will be stored in appropriate temperature and storage conditions before they are transported to Sunnybrook - where the specimens will be stored long-term. Specimens that are inadequate for study because of poor cell viability or insufficient tissue will be destroyed.

Cervical and blood samples will be taken serially from patients during their regular clinic visits. Up to 20 mL of blood and plasma may be collected for research use via venipuncture. Efforts will be made to only collect the minimum volume necessary for research use. At the patient's request, the research blood volume may be further reduced. Secondly, 10 mL of cord blood will be collected after the delivery of the baby from the umbilical vein attached to the placenta. Lastly, 1-5g samples of placental villous tissue will be collected after delivery from all subjects who have consented to this. Removal of these very small amounts of tissue will not interfere with routine histopathological examination conducted in the usual clinical care of subjects. All these samples will be labelled with the appropriate study number and kept at Sunnybrook for storage. Consent for biospecimen collection will also include permission for future use of their de-identified samples in collaborative projects with other institutions. All such collaborative projects would be subject to Ethics Board consent and relevant material transfer agreements.

ELIGIBILITY:
Inclusion Criteria:

* Consenting pregnant adults (age 18-45 years) with known or suspected risk for abnormal placentation (Abnormal Placentation Group)
* Consenting pregnant adults (age 18-45 years) with low-risk pregnancies (Control Group)
* Singleton or multiple pregnancy
* Ongoing clinical care at the participating sites, with delivery at the same institution.

Exclusion Criteria:

* None

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Female, must be pregnant
Study Population: Women age 18-45 who are pregnant
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
Biomarker levels | 18 months
  Biomarkers for disease will be quantified in biospecimens.
Pathology | 9 months
  From the database, the presence or absence of perinatal pathologies recorded in the patient's medical records will be determined. These data will be compared with biomarker levels to determine if they are correlated.

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Drewlo, PhD, Principal Investigator — Sunnybrook Research Institute

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share IPD outside of the study team as per institutional REB guidelines. Any researchers wishing to access study IPD can contact the PI.